CLINICAL TRIAL: NCT02680002
Title: Randomized, Double-Blinded, Phase 2 Study to Assess Safety & Immunogenicity of Stored Inactivated Monovalent Influenza A/Vietnam/H5N1 Virus Vaccine Administered Intramuscularly at Different Dose Levels Given With & Without Stored MF59® Adjuvant
Brief Title: Assess the Safety & Immunogenicity of Stored Inactivated Influenza H5N1 Virus Vaccine Given With & Without Stored MF59 Adjuvant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BARDA CSN 15-0001
Record Dates: First submitted 2016-01-26; First posted 2016-02-11 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2019-04

CONDITIONS: A/Vietnam/H5N1 Influenza Virus
MeSH Terms: interventions — MF59 oil emulsion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 7.5 mcg H5N1 (monobulk) Plus MF59 (monobulk) (Experimental): Two 0.5-mL doses, given at Day 0 and 21 consisting of 7.5 mcg hemagglutinin (HA) antigen stored long-term as monobulk inactivated
  Interventions: Biological: 7.5 mcg H5N1 (stored as monobulk); Other: MF59 (stored as monobulk)
- 15 mcg H5N1 (monobulk) Plus MF59 (monobulk) (Experimental): Two 0.5-mL doses, given at Day 0 and 21 consisting of 15 mcg HA antigen stored long-term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored long-term as monobulk MF59 adjuvant
  Interventions: Biological: 15 mcg H5N1 (stored as monobulk); Other: MF59 (stored as monobulk)
- 7.5 mcg H5N1 (monobulk) Plus MF59 (vials) (Experimental): Two 0.5-mL doses, given at Day 0 and 21 consisting of 7.5 mcg HA antigen stored long-term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored short-term in vials as MF59 adjuvant
  Interventions: Biological: 7.5 mcg H5N1 (stored as monobulk); Other: MF59
- 15 mcg H5N1 (monobulk) Plus MF59 (vials) (Experimental): Two 0.5-mL doses, given at Day 0 and 21 consisting of 15 mcg HA antigen stored long-term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored short-term in vials as MF59 adjuvant
  Interventions: Biological: 15 mcg H5N1 (stored as monobulk); Other: MF59
- 90 mcg H5N1 (monobulk) without MF59 (Experimental): Two 1.0-mL doses at Day 0 and 21 consisting of 90 mcg HA antigen stored long-term as monobulk inactivated A/Vietnam/H5N1 antigen formulated and filled in 2015, administered without MF59
  Interventions: Biological: 90 mcg H5N1 (stored as monobulk)
- 90 mcg H5N1 (vials) without MF59 (Experimental): Two 1.0-mL doses at Day 0 and 21 consisting of 90 mcg HA antigen stored long-term in vials as inactivated A/Vietnam/H5N1 vaccine, administered without MF59
  Interventions: Biological: 90 mcg H5N1 (stored in vials)

INTERVENTIONS:
Biological: 7.5 mcg H5N1 (stored as monobulk)
  Arms: 7.5 mcg H5N1 (monobulk) Plus MF59 (monobulk); 7.5 mcg H5N1 (monobulk) Plus MF59 (vials)
Biological: 15 mcg H5N1 (stored as monobulk)
  Arms: 15 mcg H5N1 (monobulk) Plus MF59 (monobulk); 15 mcg H5N1 (monobulk) Plus MF59 (vials)
Biological: 90 mcg H5N1 (stored as monobulk)
  Arms: 90 mcg H5N1 (monobulk) without MF59
Biological: 90 mcg H5N1 (stored in vials)
  Arms: 90 mcg H5N1 (vials) without MF59
Other: MF59
  Arms: 15 mcg H5N1 (monobulk) Plus MF59 (vials); 7.5 mcg H5N1 (monobulk) Plus MF59 (vials)
Other: MF59 (stored as monobulk)
  Arms: 15 mcg H5N1 (monobulk) Plus MF59 (monobulk); 7.5 mcg H5N1 (monobulk) Plus MF59 (monobulk)

SUMMARY:
The main purpose of this study is to assess the usability of long-term stored H5N1 antigen and adjuvant. The study is designed to assist in stockpile management by assessing the safety, reactogenicity, and immunogenicity long-term stored influenza A/Vietnam/H5N1 vaccine when administered with or without MF59® adjuvant.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, Phase 2 study to assess the safety and immunogenicity of 2 doses of long-term stored inactivated monovalent influenza A/Vietnam/H5N1 virus vaccine administered intramuscularly with or without MF59 adjuvant in healthy males and nonpregnant females, aged 18 to 49 years, inclusive. This study is designed to assist in stockpile management and will assess the usability of long-term stored H5N1 antigen (ie, stored >10 years) and adjuvant (ie, stored >5 years).

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female
* Provide written informed consent prior to study-related procedures
* Stable health status
* Access to consistent and reliable means of telephone contact
* Able to understand and comply with planned study procedures
* Agree to stay in contact with site, and no plans to move from study area for study duration

Exclusion Criteria:

* Allergic to eggs, other vaccine components, or squalene-based adjuvants
* Women with positive pregnancy test within 24 hours of vaccination, or are breastfeeding
* Females of childbearing potential who refuse acceptable birth control, if sexually active, have not used birth control for 2 months prior to study entry
* Have immunosuppression or use anticancer chemotherapy or radiation therapy within preceding 36 months
* Have an active neoplastic disease or history of hematologic malignancy
* Have long term use (≥14 consecutive days) of glucocorticoids (>20 mg/day) or high-dose inhaled steroids (>800 mcg/day) within preceding 6 months
* Diagnosis of schizophrenia, bipolar disease, or major psychiatric diagnosis
* Have been hospitalized for psychiatric illness, attempted suicide or deemed danger to self or others within past 10 years

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05-13 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Radiant Research, Inc., Atlanta, Georgia
  - Clinical Research Advantage, Inc./Ridge Family Practice, Council Bluffs, Iowa
  - Johnson County Clin-Trials, Inc., Lenexa, Kansas
  - Central Kentucky Researcch Associates, Inc., Lexington, Kentucky
  - Radiant Research, Inc., Edina, Minnesota
  - Rochester Clinical Research, Inc., Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
The study results will be posted on publicly available clinical trial registers.

REFERENCES:
- [Background] Oshansky CM, Zhou J, Gao Y, Schweinle JE, Biscardi K, DeBeauchamp J, Pavetto C, Wollish A; BRITE Study Coordination Team; Webby RJ, Cioce V, Donis RO, Bright RA. Safety and immunogenicity of influenza A(H5N1) vaccine stored up to twelve years in the National Pre-Pandemic Influenza Vaccine Stockpile (NPIVS). Vaccine. 2019 Jan 14;37(3):435-443. doi: 10.1016/j.vaccine.2018.11.069. Epub 2018 Dec 12. PMID 30553570
- See also: Safety and immunogenicity of influenza A(H5N1) vaccine stored up to twelve years in the National Pre-Pandemic Influenza Vaccine Stockpile (NPIVS) — https://www.ncbi.nlm.nih.gov/pubmed/30553570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled at 6 sites in the US.
Groups:
- 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk): Two 0.5-mL doses, given at Day 0 and 21 consisting of 7.5 mcg hemagglutinin (HA) antigen stored long term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored long term as bulk MF59 adjuvant
- 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk): Two 0.5-mL doses, given at Day 0 and 21 consisting of 15 mcg HA antigen stored long term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored long term as bulk MF59 adjuvant MF59 adjuvant
- 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials): Two 0.5-mL doses, given at Day 0 and 21 consisting of 7.5 mcg HA antigen stored long term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored short term in vials as MF59 adjuvant
  7.5 mcg H5N1 (stored as monobulk)
  MF59
- 15 mcg H5N1 (Monobulk) Plus MF59 (Vials): Two 0.5-mL doses, given at Day 0 and 21 consisting of 15 mcg HA antigen stored long term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored short term in vials as MF59 adjuvant
- 90 mcg H5N1 (Monobulk) Without MF59: Two 1.0-mL doses at Day 0 and 21 consisting of 90 mcg HA antigen stored long term as monobulk inactivated A/Vietnam/H5N1 antigen formulated and filled in 2015, administered without MF59
- 90 mcg H5N1 (Vials) Without MF59: Two 1.0-mL doses at Day 0 and 21 consisting of 90 mcg HA antigen stored long term in vials as inactivated A/Vietnam/H5N1 vaccine, administered without MF59
Period: Overall Study
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Started | 71 | 70 | 70 | 71 | 70 | 70
Day 0 (Dose 1) | 70 | 70 | 70 | 71 | 70 | 68
Day 21 (Dose 2) | 63 | 68 | 65 | 69 | 65 | 63
Day 201 | 58 | 66 | 60 | 67 | 59 | 61
Completed | 58 | 66 | 60 | 67 | 59 | 61
Not Completed | 13 | 4 | 10 | 4 | 11 | 9
Not completed — Lost to Follow-up | 5 | 1 | 4 | 2 | 0 | 2
Not completed — Physician Decision | 5 | 1 | 1 | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 2
Not completed — Missed Visit 8 (Day 201) | 2 | 1 | 3 | 1 | 5 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: Number of participants receiving at least one dose (Dose 1/Day 0) of the investigational product.
Groups:
- 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk): Two 0.5-mL doses, given at Day 0 and 21 consisting of 15 mcg HA antigen stored long term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored long term as monobulk MF59 adjuvant
- 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials): Two 0.5-mL doses, given at Day 0 and 21 consisting of 7.5 mcg HA antigen stored long term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored short term in vials as MF59 adjuvant
- Total: Total of all reporting groups
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59 | Total
Number analyzed (Participants) | 70 | 70 | 70 | 71 | 70 | 68 | 419
Age, Customized [Number; unit: participants]
  18 to <30 | 16 | 18 | 11 | 17 | 21 | 15 | 98
  30 to <40 | 22 | 21 | 26 | 28 | 22 | 31 | 150
  40 to 49 | 32 | 31 | 33 | 26 | 27 | 22 | 171
Age, Customized [Mean (Standard Deviation); unit: years] | 36.7 (8.02) | 36.8 (8.47) | 38.1 (8.37) | 35.7 (8.25) | 34.9 (8.62) | 36.0 (7.60) | 36.4 (8.24)
Age, Customized [Median (Full Range); unit: years] | 38.0 [21 to 49] | 37.5 [20 to 48] | 38.5 [18 to 49] | 37.0 [18 to 48] | 37.0 [18 to 49] | 35.0 [18 to 49] | 37 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 50 | 33 | 43 | 41 | 39 | 249
  Male | 27 | 20 | 37 | 28 | 29 | 29 | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 43 | 52 | 50 | 47 | 51 | 46 | 289
  Black or African American | 27 | 14 | 18 | 22 | 17 | 18 | 116
  Asian | 0 | 1 | 1 | 0 | 0 | 1 | 3
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Multiracial | 0 | 2 | 1 | 0 | 0 | 1 | 4
  Other | 0 | 1 | 0 | 1 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 70 | 71 | 70 | 68 | 419
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 32.79 (9.29) | 30.76 (8.59) | 31.75 (8.35) | 30.50 (8.15) | 31.76 (8.13) | 31.57 (9.27) | 31.52 (8.62)
Body Mass Index (BMI) [Median (Full Range); unit: kg/m2] | 30.93 [20.23 to 63.66] | 28.95 [17.76 to 61.42] | 29.79 [17.50 to 56.96] | 28.08 [13.89 to 53.45] | 30.21 [20.33 to 54.13] | 30.84 [17.89 to 71.43] | 29.70 [17.50 to 71.43]

OUTCOME MEASURES:

1. Primary Outcome: Number of Occurences of Mild, Moderate, or Severe Solicited Local Symptoms During the 7 Days After Each Vaccination.
Description: Occurence of mild, moderate, or severe solicited local symptoms during the 7 days (Days 0 to 7) following Dose 1
Time Frame: Days 0 to 7
Population: Participants who received Dose 1 (Day 0), analyzed up to Day 7.
Measure: Number; unit: occurrences
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 70 | 70 | 70 | 71 | 70 | 68
occurrences
  Total number solicited local AEs (Adverse Events) | 34 | 41 | 34 | 34 | 28 | 33
  Total no. Mild solicited AEs | 31 | 37 | 30 | 29 | 23 | 29
  Total no. Moderate solicited AEs | 3 | 4 | 4 | 3 | 5 | 4
  Total no. Severe solicited AEs | 0 | 0 | 0 | 2 | 0 | 0

2. Primary Outcome: Number of Occurences of Mild, Moderate, or Severe Solicited Local Symptoms During the 7 Days After Each Vaccination.
Description: Occurence of mild, moderate, or severe solicited local symptoms during the 7 days (Days 21 to 28) following Dose 2
Time Frame: Days 21 to 28
Population: Participants who received Dose 2 (Day 21), analyzed up to Day 28.
Measure: Number; unit: occurrences
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 63 | 68 | 65 | 69 | 65 | 63
occurrences
  Total number solicited local AEs (Adverse Events) | 26 | 24 | 23 | 24 | 18 | 23
  Total no. Mild solicited AEs | 26 | 22 | 23 | 23 | 17 | 21
  Total no. Moderate solicited AEs | 0 | 2 | 0 | 1 | 1 | 2
  Total no. Severe solicited AEs | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With >=1 (More Than or Equal to 1) Mild, Moderate, or Severe Solicited Local Symptoms During the 7 Days After Each Vaccination.
Description: Number of participants with >=1 mild, moderate, or severe solicited local symptoms during the 7 days (Days 0 to 7) following Dose 1
Time Frame: Days 0 to 7
Population: Participants who received Dose 1 (Day 0), analyzed up to Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 70 | 70 | 70 | 71 | 70 | 68
Participants
  Total number solicited local AEs (Adverse Events) | 25 | 31 | 27 | 27 | 22 | 25
  Total no. Mild solicited local AEs | 23 | 28 | 24 | 24 | 18 | 21
  Total no. Moderate solicited local AEs | 2 | 3 | 3 | 2 | 4 | 4
  Total no. Severe solicited local AEs | 0 | 0 | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With >=1 (More Than or Equal to 1) Mild, Moderate, or Severe Solicited Local Symptoms During the 7 Days After Each Vaccination.
Description: Number of participants with >=1 mild, moderate, or severe solicited local symptoms during the 7 days (Days 21 to 29) following Dose 2
Time Frame: Days 21 to 28
Population: Participants who received Dose 2 (Day 21), analyzed up to Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 63 | 68 | 65 | 69 | 65 | 63
Participants
  Total number solicited local AEs (Adverse Events) | 20 | 20 | 17 | 21 | 17 | 21
  Total no. Mild solicited local AEs | 20 | 19 | 17 | 20 | 16 | 19
  Total no. Moderate solicited local AEs | 0 | 1 | 0 | 1 | 1 | 2
  Total no. Severe solicited local AEs | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Mild, Moderate, or Severe Solicited Systemic Reactogenicity Symptoms During the 7 Days After Each Vaccination.
Description: Number of participants with mild, moderate, or severe solicited systemic reactogenicity adverse events during the 7 days (Days 0 to 7) following Dose 1
Time Frame: Days 0 to 7
Population: Participants who received Dose 1 (Day 0), analyzed up to Day 7.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 70 | 70 | 70 | 71 | 70 | 68
participants
  Total no. solicited systemic AEs (Adverse Events) | 20 [18.4 to 40.6] | 17 [14.8 to 36.0] | 23 [22.1 to 45.1] | 24 [23.0 to 46.0] | 17 [14.8 to 36.0] | 18 [16.5 to 38.6]
  Total no. Mild solicited systemic AEs | 13 [10.3 to 29.7] | 14 [11.4 to 31.3] | 17 [14.8 to 36.0] | 19 [16.9 to 38.6] | 13 [10.3 to 29.7] | 13 [10.6 to 30.5]
  Total no. Moderate solicited systemic AEs | 7 [4.1 to 19.5] | 3 [0.9 to 12.0] | 6 [3.2 to 17.7] | 4 [1.6 to 13.8] | 4 [1.6 to 14.0] | 3 [0.9 to 12.4]
  Total no. Severe solicited systemic AEs | 0 [0.0 to 5.1] | 0 [0.0 to 5.1] | 0 [0.0 to 5.1] | 1 [0.0 to 7.6] | 0 [0.0 to 5.1] | 2 [0.4 to 10.2]

6. Primary Outcome: Number of Participants With of Mild, Moderate, or Severe Solicited Systemic Reactogenicity Symptoms During the 7 Days After Each Vaccination.
Description: Number of participants with of mild, moderate, or severe solicited systemic reactogenicity adverse events during the 7 days (Days 21 to 28) following Dose 2
Time Frame: Days 21 to 28
Population: Participants who received Dose 2 (Day 21), analyzed up to Day 28.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 63 | 38 | 65 | 59 | 65 | 63
participants
  Total no. solicited systemic AEs (Adverse Events) | 11 [9.1 to 29.1] | 10 [7.3 to 25.4] | 11 [8.8 to 28.3] | 17 [15.1 to 36.5] | 9 [6.5 to 24.7] | 9 [6.7 to 25.4]
  Total no. Mild solicited systemic AEs | 8 [5.6 to 23.5] | 10 [7.3 to 25.4] | 10 [7.6 to 26.5] | 11 [8.2 to 26.7] | 5 [2.5 to 17.0] | 9 [6.7 to 25.4]
  Total no. Moderate solicited systemic AEs | 3 [1.0 to 13.3] | 0 [0.0 to 5.3] | 1 [0.0 to 8.3] | 6 [3.3 to 18.0] | 4 [1.7 to 15.0] | 0 [0.0 to 5.7]
  Total no. Severe solicited systemic AEs | 0 [0.0 to 5.7] | 0 [0.0 to 5.7] | 0 [0.0 to 5.5] | 0 [0.0 to 5.2] | 0 [0.0 to 5.5] | 0 [0.0 to 5.7]

7. Primary Outcome: Geometric Mean Titer (GMT) of Hemagglutination Inhibition (HAI) Antibody
Description: Geometric Mean Titer (GMT) of hemagglutination inhibition (HAI) antibody against A/Vietnam/H5N1 antigen in each study group
Time Frame: 21 days after receipt of second dose of vaccine (Day 42) (plus or minus 3 days)
Population: Participants who received Dose 2 (Day 28) of vaccine, analyzed at Day 42 (plus or minus 3 days).
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titers
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 61 | 67 | 62 | 69 | 65 | 61
antibody titers | 38 [28.7 to 50.4] | 29.6 [22.6 to 38.9] | 37.4 [28.3 to 49.4] | 49.4 [37.7 to 64.8] | 19.4 [14.6 to 25.7] | 19.9 [13.9 to 28.4]

8. Primary Outcome: Geometric Mean Titer (GMT) of Hemagglutination Inhibition (HAI) Antibody
Description: as for outcome 7
Time Frame: 21 days after receipt of second dose of vaccine (Day 42) (plus or minus 3 days)
Population: Participants who received Dose 2 (Day 28) of vaccine, analyzed at Day 42 (plus or minus 3 days).
Measure: Median (Full Range); unit: antibody titers
Groups:
- 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials): Two 0.5-mL doses, given at Day 0 and 21 consisting of 7.5 mcg HA antigen stored long term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored short-term in vials as MF59 adjuvant
- 15 mcg H5N1 (Monobulk) Plus MF59 (Vials): Two 0.5-mL doses, given at Day 0 and 21 consisting of 15 mcg HA antigen stored long term as monobulk inactivated A/Vietnam/H5N1 vaccine and MF59 stored short-term in vials as MF59 adjuvant
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 61 | 67 | 62 | 69 | 65 | 61
antibody titers | 40.0 [5 to 320] | 40.0 [5 to 226] | 40.0 [5 to 453] | 56.6 [5 to 640] | 20 [5 to 640] | 14.1 [5 to 905]

9. Secondary Outcome: Number of Participants With Vaccine-associated Serious Adverse Events (SAE) or Adverse Event of Special Interests (AESI)
Description: Number of participants with vaccine-associated serious adverse events (SAE) or adverse event of special interests (AESI) and occurence of AESIs or AEs leading to study withdrawal
Time Frame: First vaccination through 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 70 | 71 | 70 | 71 | 70 | 69
Participants
  Vaccine-associated Serious Adverse Event (SAE) | 0 | 0 | 0 | 0 | 0 | 0
  Adverse Event of Special Interest (AESI) | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) or Adverse Events (AE) Leading to Study Withdrawal.
Description: Number of participants with adverse events of special interest (AESI) or adverse events (AE) leading to study withdrawal.
Time Frame: First vaccination through approximately 13 months after first vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 70 | 71 | 70 | 71 | 70 | 69
Participants
  Adverse Event of Special Interest (AESI) | 0 | 0 | 0 | 0 | 0 | 0
  Adverse Events (AE) leading to study withdrawal | 0 | 0 | 0 | 0 | 1 | 2

11. Secondary Outcome: Number of Participants With Unsolicited Adverse Events (AE)
Description: Number of participants with unsolicited adverse events (AE) through Visit 8 (Day 201)
Time Frame: Day 0 (Visit 1) through Day 201 (Visit 8)
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 70 | 71 | 70 | 71 | 70 | 69
Participants
  Any unsolicited Adverse Event (AE) | 28 | 37 | 36 | 42 | 31 | 27
  Any severe unsolicited Adverse Event (AE) | 1 | 2 | 3 | 2 | 3 | 3

12. Secondary Outcome: Frequency of Unsolicited Adverse Events (AE)
Description: Frequency of unsolicited adverse events (AE) for 21 days following Dose 1 (Days 0-21) and after Dose 2 (>21 Days)
Time Frame: 21 days following each vaccination (Days 0-21, >21 Days)
Measure: Number; unit: Unsolicited Adverse Events (AE)
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 70 | 71 | 70 | 71 | 70 | 69
Unsolicited Adverse Events (AE)
  Days 0-21 | 184 | 179 | 186 | 202 | 156 | 174
  >21 Days | 0 | 1 | 4 | 2 | 1 | 4

13. Secondary Outcome: Occurrence of Clinical Safety Laboratory AEs
Description: Occurrence of clinical safety laboratory AEs at 7 and 21 days after each vaccination
Time Frame: 7 and 21 days after each vaccination (Days 0, 7, 21, 28, and 42)
Measure: Number; unit: Clinical safety lab results reported
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 70 | 71 | 70 | 71 | 70 | 69
Clinical safety lab results reported
  Visit 1: Day 0 | 0 | 1 | 0 | 0 | 0 | 0
  Visit 3: Day 7 | 0 | 1 | 0 | 0 | 0 | 1
  Visit 4: Day 21 | 0 | 1 | 0 | 0 | 0 | 0
  Visit 6: Day 28 | 0 | 1 | 0 | 0 | 0 | 0
  Visit 7: Day 42 | 0 | 1 | 0 | 0 | 0 | 0

14. Secondary Outcome: GMT (Geometric Mean Titers) of Serum HAI (Hemagglutination Inhibition) Antibodies
Description: Overall GMTs of HAI antibodies at baseline (Day 0) and Days 21, 28 and 201
Time Frame: Day 0 (Visit 1), Day 21 (Visit 4), Day 28 (Visit 6), Day 201 (Visit 8)
Population: Population receiving Dose 1 at Day 0 (Visit 1)
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titers
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 61 | 67 | 62 | 69 | 65 | 61
antibody titers
  Visit 1: Day 0 | 5.0 [5.0 to 5.1] | 5.0 [5.0 to 5.1] | 5.4 [5.0 to 5.8] | 5.2 [4.9 to 5.6] | 5.1 [5.0 to 5.2] | 5.3 [4.9 to 5.8]
  Visit 4: Day 21 (+1 day) | 11.8 [9.0 to 15.4] | 8.6 [7.0 to 10.4] | 8.7 [6.7 to 11.4] | 14.8 [11.1 to 19.7] | 10.8 [8.0 to 14.6] | 14.1 [9.6 to 20.9]
  Visit 6: Day 28 (+1 day) | 18.4 [13.8 to 24.5] | 18.7 [14.0 to 25.0] | 17.5 [13.2 to 23.2] | 27.9 [20.5 to 37.9] | 14.0 [10.3 to 19.1] | 20.7 [14.3 to 30.0]
  Visit 8: Day 201 (plus or minus 7 days): number analyzed (Participants) | 58 | 65 | 59 | 67 | 59 | 59
  Visit 8: Day 201 (plus or minus 7 days) | 6.2 [5.3 to 7.2] | 5.4 [5.1 to 5.7] | 5.5 [5.0 to 5.9] | 5.4 [5.1 to 5.8] | 5.9 [5.1 to 6.8] | 6.9 [5.6 to 8.6]

15. Secondary Outcome: GMT (Geometric Mean Titers) of Serum Microneutralization (MN) Antibodies
Description: GMT of serum MN antibodies at baseline (Day 0) and Days 21, 28, 42 and 201
Time Frame: Day 0 (Visit 1), Day 21 (Visit 4), Day 28 (Visit 6), Day 42 (Visit 7), Day 201 (Visit 8)
Population: Population receiving Dose 1 at Day 0 (Visit 1)
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titers
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 61 | 67 | 62 | 69 | 65 | 61
antibody titers
  Visit 1: Day 0: number analyzed (Participants) | 61 | 67 | 62 | 69 | 64 | 61
  Visit 1: Day 0 | 6.1 [5.6 to 6.6] | 5.5 [5.2 to 5.8] | 5.5 [5.2 to 5.7] | 6.0 [5.6 to 6.5] | 5.4 [5.1 to 5.7] | 5.7 [5.4 to 6.1]
  Visit 4: Day 21 (+1 day) | 12.2 [9.3 to 16.1] | 8.0 [6.9 to 9.3] | 10.9 [8.4 to 14.1] | 14.2 [11.0 to 18.4] | 10.7 [8.2 to 13.8] | 15.4 [10.5 to 22.6]
  Visit 6: Day 28 (+1 day) | 24.0 [18.6 to 31.0] | 23.8 [19.1 to 29.7] | 24.9 [19.6 to 31.6] | 31.1 [24.1 to 40.2] | 16.8 [13.2 to 21.3] | 24.0 [16.9 to 34.1]
  Visit 7: Day 42 (plus or minus 3 days) | 52.2 [39.2 to 69.7] | 43.0 [33.8 to 54.7] | 58.8 [45.4 to 76.1] | 66.4 [52.3 to 84.3] | 25.0 [20.2 to 31.0] | 30.1 [22.0 to 41.3]
  Visit 8: Day 201 (plus or minus 7 days): number analyzed (Participants) | 58 | 65 | 59 | 67 | 59 | 59
  Visit 8: Day 201 (plus or minus 7 days) | 11.3 [9.1 to 14.0] | 8.8 [7.5 to 10.1] | 10.9 [8.7 to 13.5] | 9.9 [8.3 to 11.7] | 8.9 [7.3 to 10.8] | 11.0 [8.0 to 15.0]

16. Secondary Outcome: Serum HAI (Hemagglutination Inhibition) Titer of at Least 1:40
Description: Proportion of participants achieving a serum HAI titer of at least 1:40 against the A/Vietnam/H5N1 antigen
Time Frame: Days 0 (Visit 1), 21 (Visit 4, +1day), 28 (Visit 6, +1 day), 42 (Visit 7, plus or minus 3 days), and 201 (Visit 8, plus or minus 7 days)
Population: Participants who satisfied the predefined criteria for assessment.
Measure: Count of Participants; unit: Participants
Groups:
- 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk): Two 0.5-mL doses, given at Day 0 and 21 consisting of 7.5 mcg hemagglutinin (HA) antigen stored long term as monobulk inactivated A/Vietnam/G5N1 vaccine and MF59 stored long term as bulk MF59 adjuvant
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 61 | 67 | 62 | 69 | 65 | 61
Participants
  Day 0 (Visit 1): number analyzed (Participants) | 61 | 67 | 62 | 69 | 64 | 61
  Day 0 (Visit 1) | 0 | 0 | 1 | 1 | 0 | 1
  Day 21 (Visit 4, +1 day) | 13 | 6 | 9 | 18 | 12 | 16
  Day 28 (Visit 6, +1 day) | 22 | 25 | 18 | 33 | 19 | 22
  Day 42 (Visit 7, plus or minus 3 days) | 39 | 38 | 42 | 49 | 21 | 22
  Day 201 (Visit 8, plus or minus 7 days): number analyzed (Participants) | 58 | 65 | 59 | 67 | 59 | 59
  Day 201 (Visit 8, plus or minus 7 days) | 1 | 0 | 1 | 1 | 1 | 3

17. Secondary Outcome: Seroconversion Rate (SCR) for Hemagglutination Inhibition (HAI) Antibodies
Description: Defined as proportion of subjects achieving either a prevaccination HAI titer of <1:10 and postvaccination titer of at least 1:40 or a prevaccination HAI titer of at least 1:10 and a 4-fold or greater increase of HAI postvaccination antibody titers against the A/Vietnam/H5N1 antigen; if baseline HAI titer is undetectable, it will be assigned a vaue of half the lower limit of detection.
Time Frame: Days 21, 28, 42, and 201
Population: Participants who satisfied the predefined criteria
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 61 | 67 | 62 | 69 | 65 | 61
Participants
  Visit 4: Day 21 (+1 day) | 13 | 6 | 8 | 18 | 12 | 16
  Visit 6: Day 28 (+1day): number analyzed (Participants) | 61 | 67 | 62 | 69 | 64 | 61
  Visit 6: Day 28 (+1day) | 22 | 25 | 17 | 33 | 19 | 21
  Visit 7: Day 42 (plus or minus 3 days): number analyzed (Participants) | 61 | 67 | 62 | 69 | 64 | 61
  Visit 7: Day 42 (plus or minus 3 days) | 39 | 38 | 41 | 49 | 21 | 21
  Visit 8: Day 201 (plus or minus 7 days): number analyzed (Participants) | 58 | 65 | 59 | 67 | 59 | 59
  Visit 8: Day 201 (plus or minus 7 days) | 1 | 0 | 1 | 1 | 1 | 3

18. Secondary Outcome: Seroconversion Rate (SCR) for Microneutralization (MN) Antibodies
Description: Defined as proportion of subjects achieving either a prevaccination MN titer of <1:10 and postvaccination titer of at least 1:40 or a prevaccination MN titer of at least 1:10 and a 4-fold or greater increase of MN postvaccination antibody titers against the A/Vietnam/H5N1 antigen; if baseline MN titer is undetectable, it will be assigned a vaue of half the lower limit of detection.
Time Frame: Days 21, 28, 42, and 201
Population: Participants who satisfied the predefined criteria
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
Number analyzed (Participants) | 61 | 67 | 62 | 69 | 65 | 61
Participants
  Visit 4: Day 21 (+1 day): number analyzed (Participants) | 61 | 67 | 62 | 69 | 64 | 61
  Visit 4: Day 21 (+1 day) | 10 | 3 | 11 | 13 | 9 | 12
  Visit 6: Day 28 (+1day): number analyzed (Participants) | 61 | 67 | 62 | 69 | 64 | 61
  Visit 6: Day 28 (+1day) | 18 | 21 | 23 | 31 | 15 | 20
  Visit 7: Day 42 (plus or minus 3 days): number analyzed (Participants) | 61 | 67 | 62 | 69 | 64 | 61
  Visit 7: Day 42 (plus or minus 3 days) | 42 | 43 | 44 | 52 | 23 | 23
  Visit 8: Day 201 (plus or minus 7 days): number analyzed (Participants) | 58 | 65 | 59 | 67 | 59 | 59
  Visit 8: Day 201 (plus or minus 7 days) | 5 | 1 | 8 | 3 | 4 | 7

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data were collected from Visit 1 (Day 0) through Visit 7 (Day 42); Adverse Events of Special Interest (AESI) and Serious Adverse Events (SAEs) were assessed from Visit 1 (Day 0), until exit from the study, Visit 9 (Day 386). Data currently available to Visit 8 (Day 201).
Description: Subjects recorded solicited local and systemic reactions to the vaccine or adjuvant, and other unsolicited symptoms or complaints, including start and stop dates, on an 8-day diary card following each of the 2 vaccinations. Diary cards captured unsolicited AEs for 21 days after each vaccination. Regular investigator assessment at each visit, except Visit 1. Abnormal laboratory test results judged clinically significant by investigator recorded as AEs or SAEs.
Arm/Group | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) | 90 mcg H5N1 (Monobulk) Without MF59 | 90 mcg H5N1 (Vials) Without MF59
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/71 | 0/70 | 0/71 | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/71 | 3/70 | 0/71 | 1/70 | 2/69
Other Adverse Events (participants affected / at risk) | 44/70 | 49/71 | 47/70 | 57/71 | 48/70 | 47/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) (N=70) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) (N=71) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) (N=70) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) (N=71) | 90 mcg H5N1 (Monobulk) Without MF59 (N=70) | 90 mcg H5N1 (Vials) Without MF59 (N=69)
Appendicitis perforated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Joint dislocation (left hip) determined to be displaced prosthesis.
Infected skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Left foot.
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Left foot.
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Left fifth metatarsal.
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomeningocele (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pseudomeningocele diagnosed post-operatively following anterior/posterior cervical fusion with plating, and a C5-6 right hemilaminectomy.
Abdominal pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Injury resulting from motor vehicle accident.
Gastrointestinal organ contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Injury resulting from motor vehicle accident.
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Injury resulting from motor vehicle accident.
Flank pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Injury resulting from motor vehicle accident.
Acute myocardial infarction (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) (N=70) | 15 mcg H5N1 (Monobulk) Plus MF59 (Monobulk) (N=71) | 7.5 mcg H5N1 (Monobulk) Plus MF59 (Vials) (N=70) | 15 mcg H5N1 (Monobulk) Plus MF59 (Vials) (N=71) | 90 mcg H5N1 (Monobulk) Without MF59 (N=70) | 90 mcg H5N1 (Vials) Without MF59 (N=69)
Injection site pain (General disorders) | 30 (30) | 33 (33) | 29 (29) | 33 (33) | 25 (25) | 29 (29) — General disorders and administration site conditions
Fatigue (General disorders) | 14 (14) | 14 (14) | 12 (12) | 14 (14) | 11 (11) | 12 (12) — General disorders and administration site conditions
Injection site induration (General disorders) | 8 (8) | 9 (9) | 7 (7) | 4 (4) | 4 (4) | 8 (8) — General disorders and administration site conditions
Injection site erythema (General disorders) | 6 (6) | 5 (5) | 5 (5) | 3 (3) | 6 (6) | 7 (7) — General disorders and administration site conditions
Headache (Nervous system disorders) | 17 (17) | 15 (15) | 15 (15) | 22 (22) | 13 (13) | 17 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 12 (12) | 11 (11) | 13 (13) | 7 (7) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 7 (7) | 5 (5) | 7 (7) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 5 (5) | 9 (9) | 7 (7) | 6 (6) | 11 (11)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 5 (5) | 9 (9) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Protocol implied Clinical Study Report (CSR) would include Day 386 (end-of-study) data. Following start of study it was decided CSR would include data up to and including Day 201. CSR addendum will include data from Day 201-Day 386.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data and results owned by Sponsor. Results can be used by Institution for (a) internal non-commercial research, education and patient care, and (b) as required under applicable laws and regulations. Other uses require prior written consent of Sponsor.